CLINICAL TRIAL: NCT00679822
Title: The Prevalence and Risk Factors of Sleep Disordered Breathing in a Heart Failure Program
Status: Completed | Type: Observational
Sponsor: Ohio State University (Other)
Responsible Party: Principal Investigator, Rami Khayat, Associate Professor, Ohio State University
Other Study IDs: 2007H0043
Record Dates: First submitted 2008-05-15; First posted 2008-05-19 (Estimated); Last update posted 2014-02-13 (Estimated); Status verified 2014-02

CONDITIONS: Sleep Apnea; Heart Failure
Keywords: OSA; sleep apnea; heart failure; CHF; heart clinic; clinic; obstructive sleep apnea
MeSH Terms: conditions — Sleep Apnea Syndromes; Heart Failure; Sleep Apnea, Obstructive

STUDY DESIGN:
Observational Model: Case-Only
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Heart Failure: Heart Failure Out Patients at OSU

SUMMARY:
The objective of this protocol is the evaluation of our clinical screening program for sleep disorders in patients with heart failure.

These patients have very high prevalence of Sleep Disordered Breathing (SDB), including central and obstructive sleep apnea. There is also strong evidence that SDB, if unrecognized and untreated, will worsen heart failure and may leads to serious complications. Effective treatment of SDB results in improvement in heart failure and functional status. So far there are no guidelines in the area of screening in this patient population. The only test that would reliably rule out or confirm SDB is the polysomnography (PSG) this test is expensive and technically demanding. With the current approach to diagnosis and treatment of SDB, it routinely takes up to 5-6 months between the emergence of clinical suspicion of SDB and the initiation of appropriate treatment with CPAP. This delay and cost of this traditional approach, is a significant obstacle to providing highly needed care to this very vulnerable population.

In OSU we have a state of the art Heart Failure Program and a Sleep Heart program that was created to develop an approach to prompt diagnosis and treatment of SDB in our heart failure patients. We designed an algorithm that employs validated questionnaires and FDA approved devices. We need, however to validate our algorithm against the gold standard: the PSG. Furthermore, we need to analyze the prevalence and risk factors of each sleep disorder in light of the recent changes in the management of heart failure, which may have influenced the risk factors and prevalence as we knew them. This protocol includes a combination of clinically indicated procedures, and others that are repeated for validation purposes. The accumulation and analysis of data is also done for research purposes.

DETAILED DESCRIPTION:
Patients with systolic heart failure have higher prevalence of SDB than the general middle aged population [1-3]. There is strong evidence that treatment of OSA in the general population reduces fatal and non-fatal cardiovascular events[4]. In patients with underlying heart failure and OSA, treatment with CPAP improves ejection fraction and functional outcome[5]. In patients with heart failure and CSA, there is evidence of increased sympathetic activity [6], predisposition to dsyrrythmia [7] and increased mortality. However, to date systematic diagnostic approach of SDB in this vulnerable population is not part of the guidelines for management of heart failure.

In patients with heart failure, the prevalence of Obstructive Sleep Apnea (OSA) was estimated at 24-37 % and Central Sleep Apnea (CSA) at 40%. The severity of CSA is shown to be directly related to the severity of the underlying heart failure[8]. Additionally, the management of heart failure has changed significantly since these original studies, to include b-blockade, aggressive hemodynamic targets, and device therapy[9]. Taken together, these observations call into question the applicability of this previous prevalence estimate of CSA in this patient population. Indeed, recent data suggest a decline in the incidence of CSA[10, 11]. Obstructive Sleep Apnea, on the other hand, is strongly associated with obesity. The rising incidence of obesity, and its strong association with cardiovascular disease, may suggest a rise in the incidence of OSA in this patient population.

Did the recent changes in the management of heart failure change the prevalence and distribution of SDB? What is the most effective approach to diagnosis of this highly prevalent disorder in this very vulnerable patient population? A modern cost benefit analysis and comparison against the current slow inefficient and very expensive approach is needed. An approach that combines evaluation of risk factors and an abbreviated portable study may be adequate and certainly less expensive. Our program aims at providing every heart failure patient with clinically indicating and not otherwise available screening for SDB. Validated questionnaires and screening ambulatory sleep studies are provided to every patient. Additionally, this clinical operation has no risk to patients, rather a significant benefit. The sensitivity and specificity of this surveillance approach will need to be evaluated and validated. The validation operation will bring additional benefit to our future patients. The accumulation and analysis of the data will also enable us to determine the magnitude of the sleep co-morbidity in our heart failure patients and help educate clinicians who treat similar patients nationwide

ELIGIBILITY:
Inclusion Criteria:

* OSU Heart Failure Patient
* Willingness to complete survey
* Willingness to complete take home sleep study

Exclusion Criteria:

* Neurological deficit
* Less than 18yrs old

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Out-patients at OSU's Heart Failure clinics
Sampling Method: Non-Probability Sample
Enrollment: 195 (Actual)
Dates: Start 2007-06; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Validation of Inpatient Portable Sleep Study | Baseline
  Patients at risk of Sleep Disordered Breathing with heart failure are administered a portable sleep study during their hospitalization

CONTACTS AND LOCATIONS:
Overall Officials: Rami N Khayat, MD, Principal Investigator — Ohio State University
Locations (1):
- The Ohio State University, Columbus, Ohio, United States

REFERENCES:
- [Background] Young T, Palta M, Dempsey J, Skatrud J, Weber S, Badr S. The occurrence of sleep-disordered breathing among middle-aged adults. N Engl J Med. 1993 Apr 29;328(17):1230-5. doi: 10.1056/NEJM199304293281704. PMID 8464434
- [Background] Javaheri S, Parker TJ, Liming JD, Corbett WS, Nishiyama H, Wexler L, Roselle GA. Sleep apnea in 81 ambulatory male patients with stable heart failure. Types and their prevalences, consequences, and presentations. Circulation. 1998 Jun 2;97(21):2154-9. doi: 10.1161/01.cir.97.21.2154. PMID 9626176
- [Background] Sin DD, Fitzgerald F, Parker JD, Newton G, Floras JS, Bradley TD. Risk factors for central and obstructive sleep apnea in 450 men and women with congestive heart failure. Am J Respir Crit Care Med. 1999 Oct;160(4):1101-6. doi: 10.1164/ajrccm.160.4.9903020. PMID 10508793
- [Background] Marin JM, Carrizo SJ, Vicente E, Agusti AG. Long-term cardiovascular outcomes in men with obstructive sleep apnoea-hypopnoea with or without treatment with continuous positive airway pressure: an observational study. Lancet. 2005 Mar 19-25;365(9464):1046-53. doi: 10.1016/S0140-6736(05)71141-7. PMID 15781100
- [Background] Mansfield DR, Gollogly NC, Kaye DM, Richardson M, Bergin P, Naughton MT. Controlled trial of continuous positive airway pressure in obstructive sleep apnea and heart failure. Am J Respir Crit Care Med. 2004 Feb 1;169(3):361-6. doi: 10.1164/rccm.200306-752OC. Epub 2003 Nov 3. PMID 14597482
- [Background] Spaak J, Egri ZJ, Kubo T, Yu E, Ando S, Kaneko Y, Usui K, Bradley TD, Floras JS. Muscle sympathetic nerve activity during wakefulness in heart failure patients with and without sleep apnea. Hypertension. 2005 Dec;46(6):1327-32. doi: 10.1161/01.HYP.0000193497.45200.66. Epub 2005 Nov 14. PMID 16286569
- [Background] Leung RS, Huber MA, Rogge T, Maimon N, Chiu KL, Bradley TD. Association between atrial fibrillation and central sleep apnea. Sleep. 2005 Dec;28(12):1543-6. doi: 10.1093/sleep/28.12.1543. PMID 16408413
- [Background] Solin P, Bergin P, Richardson M, Kaye DM, Walters EH, Naughton MT. Influence of pulmonary capillary wedge pressure on central apnea in heart failure. Circulation. 1999 Mar 30;99(12):1574-9. doi: 10.1161/01.cir.99.12.1574. PMID 10096933
- [Background] Sinha AM, Skobel EC, Breithardt OA, Norra C, Markus KU, Breuer C, Hanrath P, Stellbrink C. Cardiac resynchronization therapy improves central sleep apnea and Cheyne-Stokes respiration in patients with chronic heart failure. J Am Coll Cardiol. 2004 Jul 7;44(1):68-71. doi: 10.1016/j.jacc.2004.03.040. PMID 15234409
- [Background] Bradley TD, Logan AG, Kimoff RJ, Series F, Morrison D, Ferguson K, Belenkie I, Pfeifer M, Fleetham J, Hanly P, Smilovitch M, Tomlinson G, Floras JS; CANPAP Investigators. Continuous positive airway pressure for central sleep apnea and heart failure. N Engl J Med. 2005 Nov 10;353(19):2025-33. doi: 10.1056/NEJMoa051001. PMID 16282177
- [Background] Tamura A, Kawano Y, Naono S, Kotoku M, Kadota J. Relationship between beta-blocker treatment and the severity of central sleep apnea in chronic heart failure. Chest. 2007 Jan;131(1):130-5. doi: 10.1378/chest.06-0919. PMID 17218566